CLINICAL TRIAL: NCT06353698
Title: The Effect of Fasting Mimicking Diet With Chemotherapy on the Number of Blasts and Platelets and Quality of Life in Patients With Acute Lymphoid Leukemia and Acute Myeloid Leukemia
Brief Title: Fasting Mimicking Diet With Chemotherapy in Patients With Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principle Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nnftri
Record Dates: First submitted 2024-02-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Fasting Mimicking Diet; Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fasting mimicking diet (Experimental): the intervention group that receive fasting mimicking diet with chemotherapy
  Interventions: Dietary Supplement: fasting mimicking diet
- control (No Intervention): the control group that receive chemotherapy without any intervention

INTERVENTIONS:
Dietary Supplement: fasting mimicking diet — Fasting mimicking diet is limited calorie diet to enhance the effectiveness of chemotherapy
  Arms: fasting mimicking diet

SUMMARY:
The goal of this clinical trial is to investigate The effect of fasting mimicking diet with chemotherapy on the number of blasts and platelets and quality of life in patients with acute lymphoid leukemia and acute myeloid leukemia.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate The effect of fasting mimicking diet with chemotherapy on the number of blasts and platelets and quality of life in patients with acute lymphoid leukemia and acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* People who have recently been diagnosed with acute leukemia pathology and have been prescribed chemotherapy

  * Willingness to cooperate
  * BMI >18.5

Exclusion Criteria:

* diabetes
* metastases to other organ
* Unwillingness to continue the study by patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Blast cell count | at 4th week
  the number of blast cell in perpheral blood
Quality of life | at the beginning and 4th week
  Measuring the quality of life using EORTC QLQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ehsan Hejazi, PhD, Principal Investigator — Beheshti University of Medical Sciences
Locations (2):
- Iran (2):
  - Azita Hekmatdoost, Tehran, Middle East
  - Ehsan Hejazi, Tehran

IPD SHARING:
Plan to Share IPD: No